CLINICAL TRIAL: NCT05263310
Title: Clinical Trial of Expanded Advance Care Planning to Address Regimen Intensity in Older Patients at High Risk for Treatment-Induced Hypoglycemia
Brief Title: Prepare for Your Diabetes Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-1635322; R01AG068133 (NIH)
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus With Hypoglycemia; Aging; Patient Activation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: pragmatic, clinical efficacy, patient-level randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: care provider will not be informed of patient status; outcomes assessor will be blinded to allocation status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video and Action Plan handout (Experimental): Patients in the intervention arm will be given access to an educational video (Prepare for Your Diabetes Care) and will be supported in viewing the video and the Action Plan handout.
  This program will provide brief education about changing risks and benefits of diabetes treatment as patients age, elicit values and preferences regarding treatment, and help direct next conversation steps with the participant's primary care provider.
  Interventions: Behavioral: Prepare for Your Diabetes Care
- Usual Care (Active Comparator): Patients in the control arm will continue with usual care and also complete baseline, 6-month, and 12-month surveys
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Prepare for Your Diabetes Care — Educational video and Action Plan handout
  Arms: Educational Video and Action Plan handout
Behavioral: Usual Care — Control arm patients will continue with usual care
  Arms: Usual Care

SUMMARY:
As adults with type 2 diabetes age, they are increasingly vulnerable to treatment-related hypoglycemia and its related complications (including hospitalization and death). This study proposes to evaluate, in a randomized clinical trial, a strategy of expanded advance care planning to support older adults in value-aligned re-assessment of diabetes treatment regimens with their primary care team. If the aims of this project are achieved and incidence of clinically-significant hypoglycemia is reduced, this Prepare for Your Diabetes web-based patient educational care strategy could be scaled and applied in a wide variety of healthcare settings and chronic conditions in which evolving risks, benefits, and consequences of treatment require re-assessment with age.

DETAILED DESCRIPTION:
In this pragmatic, clinical efficacy, parallel group randomized clinical trial, the study will enroll eligible Kaiser Permanente Northern California members (age 75 years or greater, type 2 diabetes, prescribed insulin or sulfonylureas [SUs], and last measured HbA1c <=8%). Participants randomly allocated to the intervention arm will view the Prepare for Your Diabetes Care web-based educational module that is designed to help them prepare to discuss their diabetes medication regimens with their primary care providers and receive an Action Plan handout. Participants randomly allocated to the control arm will continue with usual care. All participants will complete baseline, 6-month, and 12-month surveys. The hypothesis is that empowering high-risk patients to engage in values-based discussions about diabetes treatment intensity will result - when clinically appropriate - in decreases in diabetes regimen intensity leading to decreased incidence of hypoglycemia over the 12-month study period. If successful, this study will provide evidence to support strategies for safer treatment in older adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Type 2 diabetes with last measured HbA1c ≤ 8.0%
* Currently prescribed insulin and/or SUs
* Kaiser Permanente Northern California member

Exclusion Criteria:

* Unable to communicate in English
* Unable to provide informed consent and/or participate in informed decision making due to cognitive or communication-related deficits
* Excluded by their primary care provider

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Any incidence of hypoglycemia | 12 months after baseline date
  Any one of the following hypoglycemia event measures:
  * Self-report to survey question: Have you had three or more symptomatic hypoglycemia episodes in past 4 weeks (survey administered at month 6 and month 12)
  * Self-report to survey question: Have you had one or more severe hypoglycemia episodes in past 6 months that resulted in passing out or needing active help from someone else (survey administered at month 6 and month 12)
  * Clinical record of any emergency department or hospital admission with primary admitting diagnosis of hypoglycemia during the 12-month study period

SECONDARY OUTCOMES:
Patient-Reported Outcome: Incidence of Severe Self-Reported Hypoglycemia | Preceding 6-month period (asked 6 and 12 months after first study-related visit)]
  Patient report of any self-reported severe hypoglycemia episodes in past 6 months that resulted in passing out or needing active help from someone else
Patient-Reported Outcome: Incidence of Symptomatic Self-Reported Hypoglycemia | Preceding 1-month period (asked 6 and 12 months after first study-related visit)
  Patient report of three or more self-reported symptomatic episodes in past 4 weeks (measured at 6- and 12-months)
Patient-Reported Outcome: Problem Areas in Diabetes | 6 and 12 months following the first study-related visit
  5-item Problem Areas in Diabetes (PAID-5) + Worry about Hypoglycemia
Clinical Utilization Outcome: Hypoglycemic-related admissions to Emergency Department or Hospital | 6 and 12 months following the first study-related visit
  Hypoglycemic-related admissions in the 6 months and 12 months following the first study-related visit
Patient-Centered Outcome: RAND Patient Satisfaction Questionnaire | 6 and 12 months following the first study-related visit
  5-item RAND Patient Satisfaction Questionnaire (PSQ III)
Patient-Centered Outcome: Perceived Efficacy in Patient - Physician Interactions | 6 and 12 months following the first study-related visit
  5-item Perceived Efficacy in Patient - Physician Interactions (PEPPI) Survey Instrument
Patient-Centered Outcome: Active Patient Participation during primary care visits | 6 - 12 months following the first study-related visit
  In a subset of patients (n = 40 in each arm, total n = 80), we will audio-record a selected primary care visit. Visit transcripts will be analyzed using the Active Patient Participation Coding Scheme [Coding Instrument] and utterances per unit time [Outcome Measure] demonstrating active patient participation related to diabetes management will be compared between arms.
Medication-Related Outcome: Aggregate measure of diabetes medication deprescribing | 12 months following the first study-related visit
  Aggregate measure of diabetes medication deprescribing between baseline and 12-month follow-up, defined as any combination of:
  * Discontinuation of either insulin or SU,
  * Reduction in dose of insulin or SU,
  * Switch from a higher risk to lower risk version of insulin (e.g. from sliding scale insulin or basal-bolus insulin to twice daily basal insulin) and/or higher risk to lower risk oral medicine (e.g. switching from SU to other oral medicine less associated with hypoglycemia).

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Kaiser Permanente Northern California - Division of Research
Locations (1):
- Kaiser Permanente - Oakland Medical Center, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee AK, Mejia JJ, Ferguson C, Li BH, Grant RW, Sudore RL. Expanded care planning paradigm for older adults with type 2 diabetes: Rationale, design, and protocol of the PREPARE for Your Diabetes Care randomized trial. Contemp Clin Trials. 2025 Jun;153:107913. doi: 10.1016/j.cct.2025.107913. Epub 2025 Apr 11. PMID 40222399